CLINICAL TRIAL: NCT07237386
Title: Comparing the Ceriter Stride One, a Pressure-sensitive Smart Insole, With Gait Parameters Measured on the GRAIL in Neurological Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2025-0386
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Incomplete Spinal Cord Injury; Traumatic Brain Injury; Acquired Brain Injury
Keywords: Gait; stroke; spinal cord injury; brain injury; smart insoles; spatiotemporal
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Brain Injuries; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insoles (Experimental): This is the group wearing smart insoles, it is the only group
  Interventions: Device: Wearing smart insoles

INTERVENTIONS:
Device: Wearing smart insoles — Participants will wear Ceriter Stride One insoles during walking on an instrumented treadmill. Parameters (like stance phase duration and swing phase duration) measured by the insoles will be compared to the same parameters measured by the instrumented treadmill with accompanying 3D motion capture system.

SUMMARY:
Ceriter Stride-One soles have been available on the market for several years. One of the features of these soles is that they can measure gait parameters while patients walk around in a functional environment. This can provide a more realistic picture of gait patterns compared to measurements taken in a laboratory setting.

At UZ Ghent, we use an advanced gait lab to measure gait parameters before and after a training period on this system, the GRAIL system. We measure similar parameters to the Ceriter Stride-One soles (support phase, swing phase, pressure on the left leg and on the right leg). In this study, we would apply these insoles to patients who are tested on the GRAIL system, according to standard care, during the test in order to compare the parameters measured by the insoles and the parameters measured by the GRAIL system. This information will give us more insight into the accuracy of the data measured with these soles so that we can apply them in future studies conducted not in the gait lab but in functional environments.

Patients who are eligible for GRAIL therapy and are therefore routinely tested are patients who are admitted or undergoing outpatient rehabilitation at the rehabilitation centre of UZ Ghent after a brain injury, stroke, spinal cord injury or amputation. Given the subject of the research and the difficulty of fitting a sole into the shoe of a prosthetic leg, only people with brain and spinal cord injuries are asked to participate in the study.

Participants must be able to step onto the GRAIL treadmill with the help of one therapist and must be able to walk for at least six minutes. Participants have to weigh less than 120 kg (treadmill safety system restriction).

As standard in our setting, participants train for 5 weeks, twice a week for 30 minutes on the GRAIL treadmill. Before and after their training period, they walk on the GRAIL for about 2 minutes and we measure a number of gait parameters: speed, step width, step length, duration of the support phase and swing phase, and how much they support on their left and right legs.

Some of these parameters can also be measured by the Ceriter Stride One sole. The aim is to investigate how comparable these data are. If these data are sufficiently comparable, the soles can be used to measure the ratio of the support and swing phases during walking in everyday tasks or in environments other than a laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Persons suffering a lesion of the central nervous system (stroke, incomplete spinal cord injury, acquired brain injury) who are admitted to the rehabilitation center of the Ghent University hospital or who follow therapy at the rehabilitation center of the Ghent University hospital as outpatients.
* Patients need to be able to walk independently during at least 6 minutes without the need of an extra person (Functional ambulation category 3 or higher).

Exclusion Criteria:

* Severe orthopedic trauma or acute trauma of the lower limbs influencing walking
* body weight that exceeds 120 kg.
* severe dizziness that makes exercising in standing position impossible
* severe cardio-pulmonary disorders that require monitoring during exercising
* patients who do not understand the task that needs to be performed in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Swing phase as a percentage of the duration of one stride | Single point of assessment at inclusion
  For each leg the duration of the swing phase will be determined as a percentage of the duration of one stride. Using the GRAIL system this will be calculated as de duration between toe-off and the following heel contact of the same leg. Using the ceriter stride one insole this will be calculated by determining the toe-off and following heel contact based on a cut-off value using the pressure sensors in the insole. For both devices it will be expressed as a percentage of the duration of one stride.
Stance phase as a percentage of the duration of one stride | Single point of assessment at inclusion
  For each leg the duration of the stance phase will be determined as a percentage of the duration of one stride. Using the GRAIL system this will be calculated as de duration between heel contact and the following toe-off of the same leg. Using the ceriter stride one insole this will be calculated by determining the heel contact and following toe-off based on a cut-off value using the pressure sensors in the insole. For both devices it will be expressed as a percentage of the duration of one stride.

SECONDARY OUTCOMES:
Stance phase as a percentage of the duration of one stride after 5 weeks | Single point of assessment at 5 weeks after inclusion
  For each leg the duration of the stance phase will be determined as a percentage of the duration of one stride. Using the GRAIL system this will be calculated as de duration between heel contact and the following toe-off of the same leg. Using the ceriter stride one insole this will be calculated by determining the heel contact and following toe-off based on a cut-off value using the pressure sensors in the insole. For both devices it will be expressed as a percentage of the duration of one stride.
Swing phase as a percentage of the duration of one stride after 5 weeks | Single point of assessment at 5 weeks after inclusion
  For each leg the duration of the swing phase will be determined as a percentage of the duration of one stride. Using the GRAIL system this will be calculated as de duration between toe-off and the following heel contact of the same leg. Using the ceriter stride one insole this will be calculated by determining the toe-off and following heel contact based on a cut-off value using the pressure sensors in the insole. For both devices it will be expressed as a percentage of the duration of one stride.
Ratio of stance phase duration | Single point of assessment at inclusion
  The ratio of the stance phase duration of the paretic leg will be calculated compared to the non-paretic leg. Or if both legs are involved, the ratio of the most impaired leg on the least impaired leg. This will determine the asymmetry in stance phase duration during walking.
Ratio of stance phase duration after 5 weeks | Single point of assessment at 5 weeks after inclusion
  The ratio of the stance phase duration of the paretic leg will be calculated compared to the non-paretic leg. Or if both legs are involved, the ratio of the most impaired leg on the least impaired leg. This will determine the asymmetry in stance phase duration during walking.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No